CLINICAL TRIAL: NCT06883279
Title: Effect of Intraplexus and Extraplexus Interscalene Block Approaches on the Incidence of Rebound Pain in Arthroscopic Shoulder Surgery: A Prospective, Randomized, Double-Blind Clinical Study
Brief Title: Effect of Interscalene Block Methods on Rebound Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Rebound pain
Record Dates: First submitted 2025-03-09; First posted 2025-03-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia; Pain, Shoulder; Pain, Postoperative
Keywords: Anesthesia; Interscalene block; Rebound pain
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraplexus approach in interscalene block (Active Comparator): The block needle will be advanced from the middle scalene muscle in a posterior-anterior direction and advanced between the C5-C6 nerve roots and the injection will be performed
  Interventions: Other: Intraplexus
- Extraplexus approach in interscalene block (Active Comparator): The block needle will first be advanced above the C5 nerve root and towards the anterior part of the brachial plexus and 10 ml of local anesthetic will be injected. Then, the needle will be withdrawn to the posterior surface of the brachial plexus and 10 ml of local anesthetic will be administered.
  Interventions: Other: Extraplexus

INTERVENTIONS:
Other: Intraplexus — The block needle will be advanced from the middle scalene muscle in a posterior-anterior direction and advanced between the C5-C6 nerve roots and the injection will be performed
  Arms: Intraplexus approach in interscalene block
Other: Extraplexus — The block needle will first be advanced above the C5 nerve root and towards the anterior part of the brachial plexus and 10 ml of local anesthetic will be injected. Then, the needle will be withdrawn to the posterior surface of the brachial plexus and 10 ml of local anesthetic will be administered.
  Arms: Extraplexus approach in interscalene block

SUMMARY:
In this study, the hypothesis that local anesthesia, not directly injected into the nerve root, may reduce the incidence of rebound pain in the interscalene block with an extraplexus approach during arthroscopic shoulder surgeries will be investigated. Rebound pain is defined as a short-term but severe pain before and after the resolution of the interscalene block and will be evaluated using the Numerical Rating Scale (NRS) (NRS ≥ 7).

DETAILED DESCRIPTION:
The study will include patients aged 18-65 years, with an American Society of Anesthesiologists (ASA) physical status of I or II, scheduled for arthroscopic shoulder surgery in the lateral decubitus position, accompanied by interscalene nerve block performed by the same surgeon. Patient characteristics (age, gender, body mass index, etc.), block procedure duration, number of needle passes, onset time of sensory block, onset time of motor block, and possible complications related to the block (paresthesia, Horner's syndrome, dyspnea, hoarseness), postoperative nausea and vomiting (PONV) status, and Quality of Recovery-15 (QoR-15) scores on the preoperative first day and postoperative days 1 and 7 will be recorded. The primary outcome parameter will be the incidence of rebound pain. Rebound pain will be defined as a short-term but severe pain before and after the resolution of the interscalene block, assessed using the Numerical Rating Scale (NRS) (NRS ≥ 7). Secondary outcomes will include the number of needle passes, block application time, onset time of sensory block, onset time of motor block, intraoperative dexmedetomidine requirement, duration of block effectiveness, postoperative pain, PONV, need for rescue analgesics, incidence of paresthesia and Horner's syndrome, dyspnea, hoarseness, duration of stay in the recovery room, duration of rebound pain, and postoperative Quality of Recovery-15 (QoR-15) scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years.
* Patients with ASA physical status I or II.
* Patients planned for arthroscopic shoulder surgery in the lateral decubitus position with interscalene nerve block.

Exclusion Criteria:

* Patients who do not consent to participate in the study.
* Block failure.
* Language acquisition deficiency.
* Obesity (body mass index > 35 kg/m²).
* Diabetes.
* Psychiatric disorders.
* Central nervous system diseases.
* Vestibular diseases.
* Presence of neuropathy and paralysis.
* Pregnancy.
* Previous open shoulder surgery.
* Allergy to local anesthetics.
* Coagulopathy.
* Severe thrombocytopenia.
* Infection at the puncture site.
* Pre-existing neuropathy in the limb to be operated.
* Use of dexamethasone.
* Use of opioid and antiemetic medications before surgery.
* Severe cardiopulmonary disease.
* Low baseline oxygen saturation.
* Conditions that prevent cooperation in the postoperative period (e.g., mental retardation, delirium).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Rebound pain | 36 hours
  Pain will be evaluated using the 0-10 Numerical Rating Scale (NRS), where 0 represents no pain and 10 represents the worst possible pain. Rebound pain will be defined as a short-term but severe pain occurring before and after the resolution of the interscalene block (NRS ≥ 7).

SECONDARY OUTCOMES:
Number of needle passes | During the block procedure time
  Number of times the needle is withdrawn and reinserted
Block performance time | During the block procedure time
  Time from the placement of the block needle to the completion of local anesthetic injection (minutes)
Rescue analgesic | 36 hours
  Pain will be evaluated using the 0-10 Numerical Rating Scale (NRS), where 0 represents no pain and 10 represents the worst possible pain. During the postoperative period, if NRS ≥ 4 occurs, 100 mg of tramadol will be administered intravenously. This situation will be defined as the need for rescue analgesia.
Duration of rebound pain | 36 hours
  Pain will be evaluated using the 0-10 Numerical Rating Scale (NRS), where 0 represents no pain and 10 represents the worst possible pain. Rebound pain will be defined as a short-term but severe pain occurring before and after the resolution of the interscalene block (NRS ≥ 7). The duration of rebound pain experienced by patients will be recorded in minutes based on the time the pain started and ended, as assessed in a questionnaire directed at the patients.
Onset of sensory block | Preoperative time
  Duration (minutes) during which there is touch sensation but no pain in the relevant dermatomal areas in the Pin-Prick test.
Onset of motor block | Preoperative time
  Duration (minutes) during which motor strength is reduced, but the arm is still movable.
Duration of block effectiveness | 36 hours
  Time (minutes) until the patient reports a significant increase in pain after the block.
PONV | 36 hours
  Significant nausea, vomiting, and/or need for rescue antiemetics.
Paresthesia | During the block procedure time
  Observations during the block procedure of 'needle prick, tingling, or electric shock radiating to the arm
Horner's syndrome | Perioperative/Periprocedural
  Miosis and ptosis of the ipsilateral pupil during the perioperative period.
Dyspnea | Perioperative/Periprocedural
  Breathing difficulty as described by the patient during the perioperative period.
Hoarseness | Perioperative/Periprocedural
  Voice changes described by the patient during the perioperative period.
Intraoperative use of dexmedetomidine | Intraoperative time
  Ramsey Sedation Scale is a tool used to assess the sedation levels of patients, and it scores from 1 to 6. A score of 1 indicates that the patient is awake, agitated, and very active; a score of 2 indicates that the patient is awake but slightly agitated. A score of 3 indicates that the patient is awake but calm, while a score of 4 indicates that the patient responds but has decreased alertness. A score of 5 indicates that the patient is not awake but responds to stimulation; a score of 6 indicates that the patient is not awake and does not respond to stimuli. In the study, the necessary amount of dexmedetomidine (μg) will be recorded for patients to fall within the 3-4 range on the Ramsey Sedation Scale.
Pain scores | 36 hours
  Evaluated using a 0-10 Numerical Rating Scale (NRS), where zero represents no pain and ten represents the worst pain imaginable.
Duration of stay in the recovery room | up to 2 hours post surgery
  Time from arrival in the recovery room to the point when discharge criteria are met
Quality of recovery | Preoperative day 1, postoperative days 1 and 7.
  The Quality of Recovery-15 (QoR-15) questionnaire consists of 15 questions rated on a scale of 0-10, with a total score evaluated out of 150. Results are classified as 'excellent' for scores above 135, 'good' for scores between 122-135, 'moderate' for scores between 90-121, and 'poor' for scores below 90.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No